CLINICAL TRIAL: NCT07344766
Title: Pilot Prolonged Exposure Teletherapy Treatment Trial for Psychogenic Nonepileptic Seizures (PNES) and Post-traumatic Stress Disorder (PTSD): A Randomized Clinical Trial
Brief Title: Treatment for Psychogenic Nonepileptic Seizures and Post-traumatic Stress Disorder Using Prolonged Exposure Therapy (PE) or Psychoeducation for PNES
Acronym: PNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast Regional Epilepsy Group (Other)
Responsible Party: Principal Investigator, Dr. Lorna Myers, Director, PNES Program, Northeast Regional Epilepsy Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCGIRB 1280734
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Psychogenic Nonepileptic Seizures (PNESs); Post Traumatic Stress Disorder PTSD
Keywords: Psychotherapy; functional dissociative seizures; nonepileptic seizures; psychogenic nonepileptic seizures
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Combat Disorders; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged exposure (Active Comparator)
  Interventions: Behavioral: imaginal and in vivo exposure
- Psychoeducational Intervention for PNES (Active Comparator): This psychoeducational treatment was based on a similar intervention reported in 2004
  Interventions: Behavioral: psychoeducation for psychogenic nonepileptic seizures

INTERVENTIONS:
Behavioral: imaginal and in vivo exposure — Prolonged exposure is a form of cognitive behavioral treatment that uses exposure to avoided memories and reminders
  Arms: Prolonged exposure
Behavioral: psychoeducation for psychogenic nonepileptic seizures — A combination of psychoeducation about PNES and skills for emotional regulation and relaxation.
  Other Names: PsychoEd for PNES
  Arms: Psychoeducational Intervention for PNES

SUMMARY:
An outpatient randomized controlled clinical trial conducted at the Northeast Regional Epilepsy Group's PNES Program, involving mental health clinicians certified in PE and trained in administering PsychoEd.

DETAILED DESCRIPTION:
A randomized parallel group trial was utilized to compare two therapeutic interventions for PNES, PE or PsychoEd, both delivered remotely via teletherapy. Each psychotherapeutic modality provided 12, 90-minute sessions. Seizure frequency was the primary outcome measure. Secondary outcome measures were depression (Beck Depression Inventory) and post-traumatic stress symptomatology (Post-Traumatic Disorder Diagnostic Scale and PTSD Checklist). Data was collected prospectively, including baseline measures before initiating treatment, upon treatment completion, and at follow-up intervals of 3, 6, and 12-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

English-speaking adults (18 years and older) Confirmed diagnosis of PNES through video-EEG monitoring Confirmed diagnosis of current PTSD At least one psychogenic non-epileptic seizure in the month prior to beginning treatment.

Exclusion Criteria:

Concurrent mixed epilepsy and PNES or video EEG findings that cannot clearly distinguish epilepsy and PNES Active suicidality Active psychotic symptoms Active substance or alcohol use or dependence that could interfere with participation in therapy Application for disability

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Nonepileptic seizure frequency | From enrollment until session 12 and at 3, 6 and 12month follow up
  frequency of nonepileptic seizures (PNES) per month

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | From enrollment to session 12 and at 3, 6 and 12 months follow up
  Self-report inventory of depressive symptoms 0-13: minimal depression, 14-19: mild, 20-28: moderate, 29-63: severe
Posttraumatic Stress Disorder Checklist (PCL) for DSM 5 | From enrollment until session 12 of treatment and at 3, 6 and 12 months follow up
  Post traumatic stress symptom checklist scores range from 0-80, higher score means worse outcome
Posttraumatic Diagnostic Scale | From enrollment until session 12 of treatment and at 3, 6 and 12 months follow up
  post traumatic diagnostic scale 0: No symptoms, 1-10: Mild symptoms, 11-20: Moderate symptoms, 21-35: Moderate to severe symptoms, >36: Severe symptoms.
Clinician Administered PTSD Scale for DSM 5 (CAPS) | From enrollment through session 12 of treatment and at 3, 6 and 12 months follow up
  Clinician-Administered PTSD Scale for DSM 5. Severity rating: 0: absent, 1: mild, 2: moderate, 3: severe, 4: extreme

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Myers, Ph.D., Principal Investigator — NEREG
Locations (1):
- Northeast Regional Epilepsy Group, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and data collected over the duration of the study.
Supporting Information: Study Protocol, ICF
Time Frame: upon completion of final data analysis until indefinitely.
Access Criteria: Qualified researchers will have access to de-identified IPD, protocol, informed consent) via online data repository
URL: https://support.dataverse.harvard.edu/

REFERENCES:
- [Background] Myers L, Vaidya-Mathur U, Lancman M. Prolonged exposure therapy for the treatment of patients diagnosed with psychogenic non-epileptic seizures (PNES) and post-traumatic stress disorder (PTSD). Epilepsy Behav. 2017 Jan;66:86-92. doi: 10.1016/j.yebeh.2016.10.019. Epub 2016 Dec 27. PMID 28038392
- [Background] Zaroff CM, Myers L, Barr WB, Luciano D, Devinsky O. Group psychoeducation as treatment for psychological nonepileptic seizures. Epilepsy Behav. 2004 Aug;5(4):587-92. doi: 10.1016/j.yebeh.2004.03.005. PMID 15256198